CLINICAL TRIAL: NCT04192344
Title: A Phase 1, Open-Label Study of ABSK021 to Assess Safety, Tolerability, and Pharmacokinetics in Patients With Advanced Solid Tumor
Brief Title: A Study to Assess the Safety, Tolerability, and Pharmacokinetics of ABSK-021 in Patients With Advanced Solid Tumor
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Abbisko Therapeutics Co, Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ABSK021-101
Record Dates: First submitted 2019-11-27; First posted 2019-12-10 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2024-08

CONDITIONS: Neoplasms; Tenosynovial Giant Cell Tumor
Keywords: Tenosynovial Giant Cell Tumor; TGCT; Solid tumors
MeSH Terms: conditions — Neoplasms; Giant Cell Tumor of Tendon Sheath

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- ABSK021 (Experimental): Dose escalation of oral ABSK021 with a starting dose of 25mg once daily will be guided by"3+3" escalation rules based on safety data until an MTD has been identified or a RDE. For each dose, patients will first receive a single dose ABSK021 tablet(s) by mouth at Day -3 and be followed by a 3-day off as a run-in period to access the safety and PK of single-dose. Then, patients will continuously receive ABSK021 once daily (QD) in repeated 28-day cycles.
  Interventions: Drug: ABSK021

INTERVENTIONS:
Drug: ABSK021 — ABSK021 oral capsule

SUMMARY:
This is an open-label phase 1 study to determine the safety and tolebility of oral ABSK021 in patients with advanced solid tumor as well as the Recommended Phase 2 dose (RP2D) of oral ABSK021. Preliminary antitumor activity will also be assessed.

DETAILED DESCRIPTION:
The study will start with a dose escalation part of single-agent ABSK021 administered in repeated 28-day cycles in patients with advanced solid for safety and tolerability. The expansion part of oral ABSK021 at recommended dose of expansion (RDE) will be followed for further evaluating safety and tolerability among selected tumor types. Preliminary antitumor activity will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed solid tumors that have progressed on or intolerant to standard therapy or whom no standard therapy exists
* ECOG (electrocorticogram) performance status 0~1
* Life expectancy ≥ 3 months
* Adequate organ function and bone marrow function

For patients with tenosynovial giant cell tumor (TGCT) :

1. A diagnosis of TGCT [i ncluding pigmented villonodular synovitis (PVNS) or giant cell tumors of the tendon sheath (GCT TS) (i) that has been histologically confirmed either by a pathologist at the treating institution or a central pathologist, and (ii) where surgical resection would be associated with potentially worsening functional limitation or severe morbidity (locally advanced disease), with morbidity determined consensually by qualified personnel (eg, two surgeons or a multi disciplinary tumor board);
2. Measurable disease as defined by RECIST 1.1 (except that a minimal size of 2 cm is required), assessed from MRI scans;
3. Others

Exclusion Criteria:

* Known allergy or hypersensitivity to any component of the investigational drug product Previous treatment with CSF-1(colony stimulating factor 1)/CSF-1R (colony stimulating factor 1 receptor) pathway inhibitors
* Known additional malignancy that is progressing or required active treatment within 3 years of the first dose of study treatment
* Inability to take oral medication or significant nausea and vomiting, malabsorption, external biliary shunt, or significant bowel resection that would preclude adequate absorption of oral medication
* Previous anti-cancer therapy, including chemotherapy, radiotherapy, endocrine therapy or molecular targeted therapy within ≤ 5-halflife or ≤ 4 weeks (whichever is shorter) prior to initiation of study treatment (chemotherapy with nitrosourea or mitomycin should be 6 weeks prior to initiation of study treatment)
* Major surgery within 4 weeks of the first dose of study drug and all surgical wounds must be healed and free of infection or dehiscence
* Prior toxicities from chemotherapy, radiotherapy, and other anti-cancer therapies, including immunotherapy that have not regressed to Grade ≤2 severity (CTCAE v5.0) with the exception of alopecia and vitiligo
* Prior corticosteroids as anti-cancer therapy within a minimum of 2 weeks of the first dose of study drug
* Concomitant use of strong inhibitors or inducers of CYP3A4
* Active central nervous system (CNS) metastases
* Impaired cardiac function or clinically significant cardiac disease
* Patients with Gilbert's Syndrome or other underlying conditions that may lead to a greater likelihood of developing LFT(liver function test) abnormalities during the study
* Known human immunodeficiency virus or active hepatitis B, or active hepatitis C infection
* Refractory/uncontrolled ascites or pleural effusion
* Pregnant or nursing

For patients with tenosynovial giant cell tumor (TGCT) :

1. Known allergy or hypersensitivity to any component of the investigational drug product
2. For expansion part, previous treatment with CSF 1/CSF 1R pathway inhibitors (not applicable for TGCT patients in US）
3. Others

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 276 (Estimated)
Dates: Start 2020-01-20 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of DLTs | At the end of Cycle 1 (each cycle is 28 days)
  DLT(dose-limiting toxicity)
Incidence and Severity of AEs | Through study completion, an average of 6 months
  Adverse events (AEs), adverse events of special interest (AESIs) and serious adverse events (SAEs)

SECONDARY OUTCOMES:
PFS | From date of enrollment until the date of first documented progression or death, assessed up to 12 months
  Progression-Free Survival (PFS)
DoR | From date of enrollment until the date of first documented progression or death, assessed up to 12 months
  Duration of Response (DoR)
DCR | 24 weeks post-dose
  Disease Control Rate (DCR)
Cmax | Pre-dose and multiple timepoints (up to 72 hours) post-dose
  The peak plasma concentration of a drug after administration
tmax | Pre-dose and multiple timepoints (up to 72 hours) post-dose
  Time to reach Cmax
Bioavailability | Pre-dose and multiple timepoints (up to 72 hours) post-dose
  The systemically available fraction of a drug
Elimination half-life | Pre-dose and multiple timepoints (up to 72 hours) post-dose
  The time required for the concentration of the drug to reach half of its original value

CONTACTS AND LOCATIONS:
Overall Officials: Siqing Fu, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (17):
- United States (4):
  - Precision NextGen Oncology, Beverly Hills, California
  - SCRI at HealthOne, Denver, Colorado
  - The Winship Cancer Institute of Emory University, Atlanta, Georgia
  - MD Anderson Cancer Center, Houston, Texas
- China (13):
  - Beijing Jishuitan Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Sun Yat-sen University, Guangdong, Guangzhou
  - Hebei Medical University Third Hospital, Shijiazhuang, Hebei
  - Henan Cancer Hospital, Zhengzhou, Henan
  - The First Affiliated Hospital of Zhengzhou Universtity, Zhengzhou, Henan
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - Nanjing Drum Tower Hospital, Nanjing, Jiangsu
  - Liaoning Cancer Hospital, Shenyang, Liaoning
  - Huashan Hospital of Fudan University, Shanghai, Shanghai Municipality
  - Shanghai Sixth People's Hospital, Shanghai, Shanghai Municipality
  - Xi'an Hong Hui Hospital, Xian, Shanxi
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - The Second Affiliated Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang